CLINICAL TRIAL: NCT02364466
Title: Multicenter Prospective Cohort Study of Peripheral T Cell Lymphoma
Brief Title: Cohort of Peripheral T Cell Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Kosin University Gospel Hospital (Other); Dankook University (Other); Soonchunhyang University Hospital (Other); Ajou University School of Medicine (Other); Yeungnam University Hospital (Other); Ulsan University Hospital (Other); Inje University (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Hallym University Medical Center (Other); Hanyang University Seoul Hospital (Other); Seoul National University Hospital (Other); Pusan National University Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); Hanyang University (Other)
Responsible Party: Principal Investigator, Sujin Kang, CRA, Korea Cancer Center Hospital
Other Study IDs: Giraffe-T
Record Dates: First submitted 2015-02-02; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Lymphoma, T-Cell, Peripheral; Febrile Neutropenia
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2019 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, observational cohort study of peripheral T cell lymphoma. Purpose is to investigate the complication including febrile neutropenia in the era of pegylated G-CSF prophylaxis.

DETAILED DESCRIPTION:
Prospective evaluation of frequencies of febrile neutropenia or infectious complications in a homogeneous population of patients with peripheral T cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naive peripheral T cell lymphoma

   Subtypes are as followings:

   Anaplastic large cell lymphoma angioimmunoblastic T cell lymphoma Peripheral T cell lymphoma-NOS Enteropathy-associated T cell lymphoma Hepatosplenic T-cell lymphoma Subcutaneous panniculitis-like T-cell lymphoma Primary cutaneous gamma-delta T-cell lymphoma Primary cutaneous CD8+ aggressive epidermotropic lymphoma
2. Scheduled to receive chemotherapy of curative intent
3. 19 years old or over
4. Expected survival is more than 6 months
5. Informed consent

Exclusion Criteria:

1. Other histology than those described above

   * Extranodal NK/T cell lymphoma
   * Other than peripheral T cell lymphoma
2. Other combined malignancy
3. Previous history of chemotherapy or radiation therapy
4. No informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peripheral T-cell lymphoma as followings:
  Anaplastic large cell lymphoma angioimmunoblastic T cell lymphoma Peripheral T cell lymphoma-NOS Enteropathy-associated T cell lymphoma Hepatosplenic T-cell lymphoma Subcutaneous panniculitis-like T-cell lymphoma Primary cutaneous gamma-delta T-cell lymphoma Primary cutaneous CD8+ aggressive epidermotropic lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Febrile neutropenia | 2 years after the last enrollment
  Incidence and severity of febrile neutropenia

SECONDARY OUTCOMES:
Infectious complication | 2 years after the last enrollment
  incidence, severity, microbiology of infection

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (18):
- South Korea (18):
  - Dankook University Hospital, Cheonan
  - Keimyung University Dongsan Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Hanyang University Guri Hospital, Guri-si
  - Inje University Ilsan Paik Hospital, Ilsan
  - National Health and Insurance Service Ilsan Hospital, Ilsan
  - Kosin Universithy Gospel Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Korea Cancer Center Hospital, Seoul
  - Asan Medical Center, Seoul
  - Choong Ang University Hospital, Seoul
  - Hallym University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan